CLINICAL TRIAL: NCT00716924
Title: Clopidogrel 600 mg and 300 mg as a Loading Dose Prior to Percutaneous Coronary Intervention And Serum Troponin Level Elevation: A Pilot Study
Brief Title: CASTLE (Clopidogrel And Serum Troponin Level Elevation)
Acronym: CASTLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9317
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 300-mg loading dose of clopidogrel given ≥ 6 and ≤ 24 hours before PCI
  Interventions: Drug: Clopidogrel
- 2 (Experimental): 600-mg loading dose of clopidogrel given ≥ 6 hours and ≤ 24 before PCI.
  Interventions: Drug: Clopidogrel
- 3 (Experimental): 600-mg loading dose of clopidogrel given immediately (≤ 45 minutes) before PCI.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 300 mg
  Arms: 1
Drug: Clopidogrel — 600 mg
  Arms: 2; 3

SUMMARY:
Primary Objective: To test if 600 mg of clopidogrel loading dose administered ≥ 6 and ≤ 24 hours prior to PCI produce a greater decrease of periprocedural release of biochemical markers (CK, CK-MB, and troponin-T and/or I) of myocardial necrosis, compared to 300 mg loading dose, given ≥ 6 and ≤ 24 hours prior to PCI or 600 mg loading dose of clopidogrel, administered immediately (≤ 45 minutes) before PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients having symptomatic coronary artery disease with objective evidence of ischemia (eg, symptoms of angina pectoris, positive stress test results or dynamic electrocardiographic (ECG) changes).
* Patients undergoing stent implantation

Exclusion Criteria:

* Any known contraindication to the use of aspirin or clopidogrel.
* Patients receiving clopidogrel within 10 days, thrombolytics within 24 hours or receiving oral anticoagulation therapy
* Elective administration of IIb/IIIa inhibitors.
* Cardiogenic shock
* Acute MI< 24 hours
* BP systolic <100 mmHg
* Left ventricular ejection fraction < 30%
* Heart failure, NYHA class III or IV
* Severe renal insufficiency (creatinine > 3.0 mg/dL)
* Platelet count <100,000/mm³
* Target lesion in a venous bypass graft
* Target lesion in a chronic occlusion

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2004-05; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Incidence of post-percutaneous coronary intervention elevation of troponin T. | At 6 and 12 months post-PCI

SECONDARY OUTCOMES:
Adverse events. | From the beginning to the end of the study
Standard hematology and blood chemistry. | At 6 and 12 months post-PCI

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Md, Study Director — Sanofi
Locations (1):
- Sanofi aventis administrative office, México, Mexico